CLINICAL TRIAL: NCT04191096
Title: A Phase 3, Randomized, Double-blind Trial of Pembrolizumab (MK-3475) Plus Enzalutamide Plus ADT Versus Placebo Plus Enzalutamide Plus ADT in Participants With Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) (KEYNOTE-991)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) Plus Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus Enzalutamide Plus ADT in Participants With Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) (MK-3475-991/KEYNOTE-991)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-991; MK-3475-991 (Other: MSD); KEYNOTE-991 (Other: MSD); jRCT2080225171 (Registry Identifier: jRCT); 2023-507024-24-00 (Registry Identifier: EU CT); U1111-1294-9592 (Registry Identifier: UTN); 2019-003633-41 (EudraCT Number)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enzalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Enzalutamide + ADT (Experimental): Starting on Day 1 of each 21-day cycle, participants receive 200 mg pembrolizumab IV every 3 weeks (Q3W) for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily, while maintaining continuous ADT with a luteinizing-hormone releasing hormone (LHRH) agonist or antagonist during study treatment. Participants will continue to receive enzalutamide and ADT until criteria for discontinuation are met.
  Interventions: Biological: Pembrolizumab; Drug: Enzalutamide; Drug: Androgen Deprivation Therapy (ADT)
- Placebo + Enzalutamide + ADT (Placebo Comparator): Starting on Day 1 of each 21-day cycle, participants receive placebo IV Q3W for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily, while maintaining continuous ADT with a LHRH agonist or antagonist during study treatment. Participants will continue to receive enzalutamide and ADT until criteria for discontinuation are met.
  Interventions: Drug: Enzalutamide; Drug: Androgen Deprivation Therapy (ADT); Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab is administered as an IV infusion at 200 mg on Day 1 of each 21-day cycle for up to 35 cycles.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Enzalutamide + ADT
Drug: Enzalutamide — Enzalutamide is administered orally as capsules/tablets at a dosage of 160 mg daily. Enzalutamide is administered continuously until criteria for discontinuation are met.
  Other Names: XTANDI®
Drug: Androgen Deprivation Therapy (ADT) — Stable regimen of ADT (LHRH agonist or antagonist) at a dose and frequency of administration that is consistent with the local product label.
Other: Placebo — Placebo infusion solution is administered as an IV infusion on Day 1 of each 21-day cycle for up to 35 cycles.
  Arms: Placebo + Enzalutamide + ADT

SUMMARY:
This study will assess the efficacy and safety of pembrolizumab plus enzalutamide plus Androgen Deprivation Therapy (ADT) versus placebo plus enzalutamide plus ADT in participants with mHSPC. The primary hypothesis is that in participants with mHSPC, the combination of pembrolizumab plus enzalutamide plus ADT is superior to placebo plus enzalutamide plus ADT with respect to 1) radiographic progression-free survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR) and 2) overall survival (OS). As of 19-JAN-2023, the study was unblinded and all study participants stopped ongoing treatment with pembrolizumab/placebo and will continue to receive Standard of Care treatment until meeting protocol-specified discontinuation criteria if deriving clinical benefit. Safety analysis will be performed at the end of the study; there will be no further analyses for efficacy and electronic patient-reported outcome (ePRO) endpoints collected from participants beyond the IA1 cutoff date. All study participants will stop ongoing treatment with pembrolizumab/placebo. Exceptions may be requested for study participants who, in the assessment of their study physician, are benefitting from the combination of enzalutamide and pembrolizumab, after consulting with the Sponsor. All other study participants should be discontinued from study and be offered standard of care (SOC) treatment as deemed necessary by the Investigator. If enzalutamide as SOC is not accessible off study to the participant, central sourcing may continue. As of Amendment 04, disease progression will no longer be centrally verified, participants will only be assessed locally. As of Amendment 4, Second Course treatment is not an option for participants. There are currently no participants in the Second Course Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male participants with histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has metastatic disease assessed by investigator and verified by BICR by either ≥2 bone lesions on bone scan and/or visceral disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Willing to maintain continuous Androgen Deprivation Therapy (ADT) with a luteinizing-hormone releasing hormone (LHRH) agonists or antagonists during study treatment or have a history of bilateral orchiectomy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 10 days of randomization
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses prior to randomization
* Has adequate organ function
* Has provided newly obtained core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed). Participants with bone only or bone predominant disease may provide a bone biopsy sample
* Male participants must agree to the following during the intervention period and for at least 120 days after the last dose of study intervention: Refrain from donating sperm PLUS either be abstinent from heterosexual intercourse and agree to remain abstinent OR agree to use contraception, unless confirmed to be azoospermic
* Male participants must agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to randomization and not recovered adequately from the toxicities and/or complications
* Has a gastrointestinal disorder affecting absorption or is unable to swallow tablets/capsules
* Has an active infection (including tuberculosis) requiring systemic therapy
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has known active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has known or suspected central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of seizure or any condition that may predispose to seizure
* Has a history of loss of consciousness within 12 months of screening
* Has had myocardial infarction or uncontrolled angina within 6 months prior to randomization, or has New York Heart Association class III or IV congestive heart failure or a history of New York Heart Association class III or IV congestive heart failure
* Has hypotension (systolic blood pressure <86 millimeters of mercury [mmHg]) or uncontrolled hypertension (systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg) at the screening visit
* Has a history of clinically significant ventricular arrhythmias
* Has hypersensitivity to pembrolizumab and/or enzalutamide and/or any of their excipients
* Has received prior ADT as neoadjuvant/adjuvant therapy for non-metastatic prostate cancer for >39 months in duration or within 9 months prior to randomization or with evidence of disease progression while receiving ADT
* Has had prior treatment with a next generation hormonal agent (eg, abiraterone, enzalutamide, apalutamide, darolutamide)
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received a live vaccine within 30 days prior to randomization
* Has a "superscan" bone scan
* Has had an allogenic tissue/solid organ transplant
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has received any prior pharmacotherapy, radiation therapy or surgery for metastatic prostate cancer with the following exceptions:

  1. Up to 3 months of ADT or orchiectomy with or without concurrent first-generation antiandrogens, if patient was not treated with docetaxel
  2. May have 1 course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 4 weeks prior to randomization
  3. For participants with low volume metastatic disease, may have 1 course of definitive radiotherapy if it was administered at least 4 weeks prior to randomization
  4. Up to 6 cycles of docetaxel therapy with final treatment administration completed within 2 months of randomization and no evidence of disease progression. In these participants up to 6 months of ADT permitted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1251 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2026-02-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (234):
- United States (27):
  - Alaska Clinical Research Center ( Site 0274), Anchorage, Alaska
  - Providence Alaska Medical Center ( Site 0276), Anchorage, Alaska
  - City of Hope Medical Center ( Site 0217), Duarte, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0241), Los Angeles, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 0236), Aurora, Colorado
  - Hartford HealthCare Medical Group ( Site 0212), Manchester, Connecticut
  - Smilow Cancer Center at Yale-New Haven ( Site 0250), New Haven, Connecticut
  - Sibley Memorial Hospital ( Site 0275), Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University ( Site 0209), Atlanta, Georgia
  - The University of Chicago ( Site 0264), Chicago, Illinois
  - Springfield Clinic [Springfield, IL] ( Site 0240), Springfield, Illinois
  - Cotton-O'Neil Cancer Center ( Site 0228), Topeka, Kansas
  - The Sidney Kimmel Comprehensive Cancer Center ( Site 0204), Baltimore, Maryland
  - St. Vincent Frontier Cancer Center-Research ( Site 0213), Billings, Montana
  - Comprehensive Cancer Centers of Nevada ( Site 0269), Las Vegas, Nevada
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0270), New York, New York
  - Weill Cornell Medical College ( Site 0263), New York, New York
  - Associated Medical Professionals of NY ( Site 0251), Syracuse, New York
  - Duke University ( Site 0206), Durham, North Carolina
  - TriState Urologic Services PSC Inc. dba The Urology Group ( Site 0253), Cincinnati, Ohio
  - MidLantic Urology ( Site 0273), Bala-Cynwyd, Pennsylvania
  - Ralph H. Johnson VA Center ( Site 0256), Charleston, South Carolina
  - Carolina Urologic Research Center ( Site 0259), Myrtle Beach, South Carolina
  - Urology Associates [Nashville, TN] ( Site 0233), Nashville, Tennessee
  - Inova Health System ( Site 0205), Fairfax, Virginia
  - Urology of Virginia ( Site 0224), Virginia Beach, Virginia
  - Fred Hutchinson Cancer Center ( Site 0258), Seattle, Washington
- Australia (9):
  - Chris OBrien Lifehouse ( Site 0300), Camperdown, New South Wales
  - Port Macquarie Base Hospital ( Site 0301), Port Macquarie, New South Wales
  - Riverina Cancer Care Center ( Site 0302), Wagga Wagga, New South Wales
  - Gallipoli Medical Research Ltd ( Site 0309), Greenslopes, Queensland
  - John Flynn Hospital & Medical Centre ( Site 0308), Tugun, Queensland
  - Box Hill Hospital ( Site 0304), Box Hill, Victoria
  - Monash Health ( Site 0305), Clayton, Victoria
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0306), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0311), Perth, Western Australia
- Austria (4):
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 0901), Linz, Upper Austria
  - Landeskrankenhaus Salzburg - Universitatklinikum der PMU ( Site 0900), Salzburg
  - Krankenhaus der Barmherzigen Brüder Wien ( Site 0904), Vienna
  - Medizinische Universität Wien ( Site 0903), Vienna
- Brazil (7):
  - Oncocentro Ceara ( Site 2309), Fortaleza, Ceará
  - Instituto de Cancer e Transplante de Curitiba ICTR ( Site 2306), Curitiba, Paraná
  - Hospital Sao Vicente de Paulo ( Site 2303), Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre ( Site 2304), Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia Reichow ( Site 2308), Blumenau, Santa Catarina
  - Fundacao Dr Amaral Carvalho ( Site 2302), Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 2305), São Paulo
- Canada (6):
  - The Ottawa Hospital ( Site 0100), Ottawa, Ontario
  - Niagara Health System - St. Catharines ( Site 0107), St. Catharines, Ontario
  - CISSS de la Monteregie-Centre ( Site 0105), Greenfield Park, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0109), Montreal, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0106), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0101), Québec, Quebec
- Chile (7):
  - IC La Serena Research ( Site 2406), La Serena, Coquimbo Region
  - Clinica Universidad Catolica del Maule ( Site 2407), Talca, Maule Region
  - Clinica Alemana ( Site 2408), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 2402), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2403), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 2401), Temuco, Región de la Araucanía
  - Oncocentro ( Site 2400), Viña del Mar, Región de Valparaíso
- China (24):
  - Peking University First Hospital ( Site 0800), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0802), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 0815), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 0816), Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University-Urology ( Site 0837), Guangdong, Guangdong
  - Sun Yat-Sen University Cancer Center ( Site 0825), Guangzhou, Guangdong
  - Sun Yat Sen Memorial Hospital ( Site 0819), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0838), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0822), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0818), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0829), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0833), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0817), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 0811), Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 0821), Nanchang, Jiangxi
  - The Second Affiliated Hosp of Xi'an Jiaotong Univ College of Medicine ( Site 0831), Xi'an, Shaanxi
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0807), Shanghai, Shanghai Municipality
  - The first affiliated Hospital of Xi an Jiaotong University ( Site 0812), Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0804), Tianjin, Tianjin Municipality
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0808), Hangzhou, Zhejiang
  - The 1st Affil Hosp of College of Medicine, Zhejiang Univ ( Site 0830), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 0809), Hangzhou, Zhejiang
  - Ningbo First Hospital-Urology ( Site 0835), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0834), Wenzhou, Zhejiang
- Colombia (5):
  - Clinica de la Costa S.A.S. ( Site 2504), Barranquilla, Atlántico
  - Administradora Country SA - Clinica del Country ( Site 2507), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia E.S.E ( Site 2506), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 2509), Valledupar, Cesar Department
  - Hemato Oncologos ( Site 2503), Cali, Valle del Cauca Department
- Denmark (5):
  - Rigshospitalet ( Site 1005), Copenhagen, Capital Region
  - Herlev og Gentofte Hospital. ( Site 1004), Herlev, Capital Region
  - Aalborg Universitetshospital ( Site 1000), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 1003), Odense, Region Syddanmark
  - Vejle Sygehus ( Site 1002), Vejle, Region Syddanmark
- Finland (4):
  - Keski-Suomen keskussairaala ( Site 1017), Jyväskylä, Central Finland
  - Tampereen yliopistollinen sairaala ( Site 1022), Tampere, Pirkanmaa
  - HYKS ( Site 1020), Helsinki, Southwest Finland
  - TYKS T-sairaala Syopatautien pkl ( Site 1019), Turku, Southwest Finland
- France (13):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 1114), Strasbourg, Alsace
  - Centre Georges Francois Leclerc ( Site 1112), Dijon, Cote-d Or
  - CHU-Jean Minjoz ( Site 1101), Besançon, Doubs
  - CHU de Brest -Site Hopital Morvan ( Site 1103), Brest, Finistere
  - Institut Bergonie ( Site 1104), Bordeaux, Gironde
  - Centre Bourgogne ( Site 1119), Lille, Hauts-de-France
  - Hopital Foch ( Site 1105), Suresnes, Hauts-de-Seine
  - C.H.R.U. de Rennes. Hopital de Pontchaillou ( Site 1117), Rennes, Ille-et-Vilaine
  - Institut Jean Godinot-Clinical Research Unit ( Site 1118), Reims, Marne
  - Centre D Oncologie de Gentilly ( Site 1107), Nancy, Meurthe-et-Moselle
  - Centre Leon-Berard ( Site 1110), Lyon, Rhone
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud ( Site 1102), Pierre-Bénite, Rhone
  - Hopital Henri Mondor ( Site 1116), Créteil, Val-de-Marne
- Germany (9):
  - Universitaetsklinikum Freiburg ( Site 1200), Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen - Grosshadern ( Site 1210), Munich, Bavaria
  - Klinikum Rechts der Isar ( Site 1206), München, Bavaria
  - Klinikum Nuernberg Nord ( Site 1213), Nuremberg, Bavaria
  - Staedtisches Klinikum Braunschweig gGmbH ( Site 1217), Braunschweig, Lower Saxony
  - Universitaetsklinikum der Technischen Universitaet Dresden ( Site 1204), Dresden, Saxony
  - Universitaetsklinikum Magdeburg A.o.R. ( Site 1211), Magdeburg, Saxony-Anhalt
  - Charite Universitaetsmedizin Berlin ( Site 1201), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 1212), Hamburg
- Ireland (6):
  - St Vincents University Hospital ( Site 1300), Dublin, Dublin
  - Cork University Hospital ( Site 1304), Cork
  - Tallaght University Hospital ( Site 1301), Dublin
  - Beaumont Hospital ( Site 1302), Dublin
  - University Hospital Limerick ( Site 1305), Limerick
  - University Hospital Waterford ( Site 1303), Waterford
- Israel (6):
  - Rambam Health Care Campus-Oncology Division ( Site 1400), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 1404), Jerusalem
  - Meir Medical Center ( Site 1401), Kfar Saba
  - Rabin Medical Center ( Site 1402), Petah Tikva
  - Sourasky Medical Center ( Site 1403), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 1405), Ẕerifin
- Italy (10):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 1503), Meldola, Forli-Cesena
  - Fondazione Policlinico Universitario A. Gemelli ( Site 1512), Rome, Lazio
  - Istituto Clinico Humanitas Research Hospital ( Site 1500), Rozzano, Lombardy
  - Centro Di Riferimento Oncologico ( Site 1511), Aviano, Pordenone
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 1509), Bari
  - Azienda Ospedaliera Cannizzaro ( Site 1501), Catania
  - Istituto Nazionale dei Tumori ( Site 1510), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1508), Napoli
  - Azienda Ospedaliera Santa Maria ( Site 1502), Terni
  - A.O. Verona-Ospedale Civile Maggiore Borgo-Trento ( Site 1504), Verona
- Japan (19):
  - Toho University Sakura Medical Center ( Site 0732), Sakura, Chiba
  - Ehime University Hospital ( Site 0745), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 0730), Sapporo, Hokkaido
  - Kitasato University Hospital ( Site 0734), Sagamihara, Kanagawa
  - Yokohama City University Medical Center ( Site 0735), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 0744), Kashihara, Nara
  - Kindai University Hospital ( Site 0743), Sayama, Osaka
  - The University of Osaka Hospital ( Site 0742), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 0737), Hidaka, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 0736), Koshigaya, Saitama
  - Hamamatsu University Hospital ( Site 0748), Hamamatsu, Shizuoka
  - Yamaguchi University Hospital ( Site 0746), Ube, Yamaguchi
  - Chiba Cancer Center ( Site 0733), Chiba
  - Harasanshin Hospital ( Site 0747), Fukuoka
  - Nagano Municipal Hospital ( Site 0731), Nagano
  - Osaka Metropolitan University Hospital ( Site 0741), Osaka
  - Toranomon Hospital ( Site 0740), Tokyo
  - Nippon Medical School Hospital ( Site 0738), Tokyo
  - Tokyo Women's Medical University ( Site 0739), Tokyo
- Mexico (6):
  - Hospital San Lucas Cardiologica del Sureste ( Site 2606), Tuxtla Gutiérrez, Chiapas
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 2607), Guadalajara, Jalisco
  - Centro Estatal de Cancerologia de Chihuahua ( Site 2608), Chihuahua City
  - Grupo Medico Camino SC ( Site 2613), Mexico City
  - Centro Oncologico Internacional. SEDNA ( Site 2609), Mexico City
  - Boca Raton Clinical Research QTO ( Site 2611), Querétaro
- Netherlands (7):
  - Radboud University Medical Center ( Site 1606), Nijmegen, Gelderland
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 1603), Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum ( Site 1601), Amsterdam, North Holland
  - Isala Klinieken, Locatie Sophia ( Site 1604), Zwolle, Overijssel
  - Franciscus Gasthuis en Vlietland ( Site 1605), Schiedam, South Holland
  - Meander Medisch Centrum ( Site 1602), Amersfoort, Utrecht
  - St. Antonius Ziekenhuis ( Site 1600), Utrecht
- Auckland City Hospital ( Site 0321), Auckland, New Zealand
- Peru (5):
  - Hospital Nacional Carlos Alberto Seguin Escobedo ESSALUD ( Site 2700), Arequipa, Ariqipa
  - Clinica Peruano Americana S.A. ( Site 2702), Trujillo, La Libertad
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 2708), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 2706), Lima
  - Hospital Militar Central [Lima, Peru] ( Site 2704), Lima
- Poland (10):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 1710), Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki nr 1 im. Dr. Antoniego Jurasza w Bydgoszczy ( Site 1720), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 1716), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 1718), Torun, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki w Krakowie ( Site 1707), Krakow, Lesser Poland Voivodeship
  - Radomskie Centrum Onkologii ( Site 1701), Radom, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1700), Przemyśl, Podkarpackie Voivodeship
  - Wojewodzki Szpital Specjalistyczny nr 4 w Bytomiu ( Site 1717), Bytom, Silesian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 1709), Koszalin, West Pomeranian Voivodeship
  - Twoja Przychodnia - Szczeciskie Centrum Medyczne ( Site 1721), Szczecin, West Pomeranian Voivodeship
- Russia (5):
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 1810), Krasnoyarsk, Krasnoyarsk Krai
  - SBIH City clinical hospital named after D.D. Pletniov ( Site 1813), Moscow, Moscow
  - Russian Scientific Center of Roentgenoradiology ( Site 1800), Moscow, Moscow
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 1805), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 1809), Omsk, Omsk Oblast
- South Korea (7):
  - Chonnam National University Hwasun Hospital ( Site 0406), Jeollanam-do, Jeonranamdo
  - National Cancer Center ( Site 0400), Gyeonggi-do, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0401), Seongnam-si, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 0404), Daegu, Kyongsangbuk-do
  - Seoul National University Hospital ( Site 0405), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0402), Seoul
  - Asan Medical Center ( Site 0403), Seoul
- Spain (7):
  - Instituto Catalan de Oncologia - ICO ( Site 1901), L'Hospitalet de Llobregat, Barcelona
  - Institut Català d'Oncologia (ICO) - Girona ( Site 1900), Girona, Gerona
  - Hospital Universitario Lucus Augusti ( Site 1905), Lugo
  - Hospital Universitario Ramon y Cajal ( Site 1902), Madrid
  - Hospital Clinico San Carlos ( Site 1906), Madrid
  - Hospital 12 de Octubre de Madrid ( Site 1903), Madrid
  - Hospital Virgen de la Macarena ( Site 1904), Seville
- Switzerland (4):
  - Kantonsspital St. Gallen ( Site 2000), Sankt Gallen, Canton of St. Gallen
  - CHUV (centre hospitalier universitaire vaudois) ( Site 2002), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 2001), Zurich, Canton of Zurich
  - Kantonsspital Graubuenden ( Site 2003), Chur, Kanton Graubünden
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital ( Site 0504), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 0503), Tainan
  - National Taiwan University Hospital ( Site 0500), Taipei
  - Taipei Veterans General Hospital ( Site 0501), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0502), Taoyuan District
- Thailand (4):
  - Chulalongkorn Hospital, Medical Oncology Unit ( Site 0600), Bangkok, Bangkok
  - Ramathibodi Hospital. ( Site 0601), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 0602), Bangkok, Bangkok
  - Srinagarind Hospital ( Site 0604), Khon Kaen
- Turkey (Türkiye) (7):
  - Ankara Bilkent Sehir Hastanesi ( Site 2103), Ankara, Adana
  - Acibadem Adana Hastanesi ( Site 2106), Adana
  - Ankara Universitesi Tip Fakultesi. ( Site 2101), Ankara
  - Hacettepe Universitesi Tıp Fakultesi ( Site 2105), Ankara
  - Istanbul Uni. Cerrahpasa Tip Fakultesi ( Site 2100), Istanbul
  - Ege University Medical Faculty Tulay Aktas Oncology Hospital ( Site 2102), Izmir
  - Konya Necmettin Erbakan University Medical Faculty ( Site 2104), Konya
- United Kingdom (5):
  - Aberdeen Royal Infirmary ( Site 1315), Aberdeen, Aberdeen City
  - Royal Cornwall Hospitals NHS Trust ( Site 1317), Truro, Cornwall
  - University College London Hospitals NHS Foundation Trust ( Site 1320), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 1318), London, London, City of
  - Velindre Cancer Centre Hospital ( Site 1322), Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Gratzke C, Kwiatkowski M, De Giorgi U, Martins da Trindade K, De Santis M, Armstrong AJ, Niu C, Liu Y, Poehlein CH. KEYNOTE-991: pembrolizumab plus enzalutamide and androgen deprivation for metastatic hormone-sensitive prostate cancer. Future Oncol. 2023 Jan 27. doi: 10.2217/fon-2022-0776. Online ahead of print. PMID 36705526
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26244&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1251 randomized participants1250 participants received treatment. The safety analyses were conducted using all participants as treated population, which included all randomized participants who received at least 1 dose of study intervention.
Groups:
- Pembrolizumab + Enzalutamide + ADT: Participants received 200 mg pembrolizumab IV on Day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally once daily (QD), while maintaining continuous ADT with a luteinizing-hormone releasing hormone (LHRH) agonist or antagonist during study treatment. Participants received enzalutamide and ADT until criteria for discontinuation were met.
- Placebo + Enzalutamide + ADT: Participants received placebo IV on Day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years), plus 160 mg enzalutamide taken orally QD, while maintaining continuous ADT with a LHRH agonist or antagonist during study treatment. Participants received enzalutamide and ADT until criteria for discontinuation are met.
Period: Overall Study
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Started | 626 | 625
Completed | 0 | 0
Not Completed | 626 | 625
Not completed — Death | 102 | 89
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Participants Ongoing | 518 | 530

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT | Total
Number analyzed (Participants) | 626 | 625 | 1251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (8.3) | 67.6 (8.2) | 67.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 626 | 625 | 1251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 112 | 231
  Not Hispanic or Latino | 505 | 510 | 1015
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 13 | 32
  Asian | 99 | 118 | 217
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 17 | 14 | 31
  White | 447 | 440 | 887
  More than one race | 39 | 37 | 76
  Unknown or Not Reported | 2 | 2 | 4
Prior Docetaxel for Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) at Baseline [Count of Participants; unit: Participants] — Prior docetaxel usage was defined as up to 6 cycles of docetaxel therapy for mHSPC as long as final treatment administration was completed within 2 months of randomization and no evidence of disease progression during or after completion of therapy was noted. mHSPC was defined as histologically or cytologically confirmed prostate adenocarcinoma without small cell histology.
  Yes= participants with confirmed prior docetaxel use at baseline.
  No = participants with no prior docetaxel usage at baseline.
  Participants
    Yes | 64 | 61 | 125
    No | 562 | 564 | 1126
Presence of High-Volume Disease at Baseline [Count of Participants; unit: Participants] — High volume disease was defined as presence of visceral metastases or ≥4 bone lesions with ≥1 beyond the vertebral bodies and pelvis.
  Yes = presence of high-volume disease at baseline. No = absence of high-volume disease at baseline.
  Participants
    Yes | 392 | 398 | 790
    No | 234 | 227 | 461

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: rPFS was defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Progression as per modified RECIST 1.1 was ≥20% increase in sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and was persistent for ≥6 weeks. The rPFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without a rPFS event were censored at the date of last disease assessment.
Time Frame: Up to approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for rPFS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for rPFS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.9467, Log Rank — A one-sided p-value was calculated using the log-rank test stratified by prior docetaxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No) with small strata; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.96 to 1.49] — HR and associated 95% Confidence Interval (CI) were calculated using Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by prior docetaxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No)

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for OS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for OS cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.85122, Log Rank — One-sided p-value based on log-rank test stratified by prior docetaxel for mHSPC (Yes vs No) and presence of high-volume disease (Yes vs No) with small strata; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.88 to 1.53] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Initiation of the First Subsequent Anti-cancer Therapy or Death (TFST)
Description: TFST was defined as the time from randomization to initiation of the first subsequent anti-cancer therapy or death; whichever occurred first. The TFST was calculated using the product limit (Kaplan-Meier) method for censored data. Participants without documented event at time of analysis will be censored at the date of last known time to have not received subsequent new anti-cancer therapy.
Time Frame: Up to Approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [29.0 to NA] — NA = Median and upper limit of 95% CI for TFST cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TFST cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.97907, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.01 to 1.54] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (TTSSRE)
Description: TTSSRE was the time from randomization to the first symptomatic skeletal-related event defined as: use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms, occurrence of new symptomatic pathologic bone fracture (vertebral or nonvertebral), occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention, whichever occurs first. The TTSSRE was calculated using the Kaplan-Meier method for censored data. Participants without symptomatic skeletal-related events were censored at the last evaluable assessment.
Time Frame: Up to Approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTSSRE cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTSSRE cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.27202, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.61 to 1.30] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was the time from randomization to PSA progression. The PSA progression date was defined as the date of 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, or 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline. Time to PSA was calculated using Kaplan-Meier method for censored data. Participants without PSA progression were censored at the last PSA date.
Time Frame: Up to Approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for Time to PSA Progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for Time to PSA Progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.2972, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.23] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Radiographic Soft Tissue Progression Per Soft Tissue Rules of PCWG-Modified RECIST 1.1 as Assessed by BICR
Description: The time to radiographic soft tissue progression was defined as the time from randomization to radiographic soft tissue progression per soft tissue rules of PCWG-modified RECIST 1.1 as assessed by BICR. Progression was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered progression. Time to radiographic soft tissue progression was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants without radiographic soft tissue progression were censored at the last evaluable assessment.
Time Frame: Up to Approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for time to radiographic soft tissue progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for time to radiographic soft tissue progression cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.6863, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.81 to 1.41] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Pain Progression (TTPP) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) Item #3 ("Worst Pain in 24 Hours") and Opiate Use
Description: TTPP was defined as the time from randomization to pain progression as determined by Item 3 of the BPI-SF. Pain progression was defined as: 1) For participants asymptomatic at baseline: a >2-point change from baseline in the average BPI-SF item 3 score at 2 consecutive visits or initiation of opioid use for pain 2) For participants symptomatic at baseline (average BPI-SF Item 3 score >0 and/or currently taking opioids; a >2-point change from baseline in the average BPI-SF Item 3 score and the average worst pain score >4 and no decrease in average opioid use. TTPP was calculated using the Kaplan-Meier method for censored data. Participants who had > 2 consecutive visits that were not evaluable for pain progression were censored at the last evaluable assessment.
Time Frame: Up to Approximately 32 months
Population: All randomized participants who received at least one dose of study treatment, and who had at least 1 BPI-SF assessment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 622 | 622
Months | NA [25.4 to NA] — NA = Median and upper limit of 95% CI for TTPP cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for TTPP cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.9235, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.95 to 1.39] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time From Randomization to Disease Progression as Determined by Investigator Assessment After Next-line of Therapy or Death From Any Cause, Whichever Occurs First (PFS2)
Description: PFS2 was defined as the time from randomization to disease progression as determined by investigator assessment of radiological or clinical progression after next-line of therapy or death from any cause, whichever occurs first.
Time Frame: Up to Approximately 32 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 626 | 625
Months | NA [29.0 to NA] — NA = Median and upper limit of 95% CI for PFS2 cannot be calculated at the time of last disease assessment due to insufficient number of participants with events | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for PFS2 cannot be calculated at the time of last disease assessment due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.8801, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.90 to 1.50] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: PSA response rate was the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by >50%. The reduction in PSA level was confirmed by an additional PSA evaluation performed >3 weeks from the original response.
Time Frame: Up to Approximately 32 Months
Population: All randomized participants who had a baseline PSA measurement and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 619 | 617
Percentage of participants | 90.3 [87.7 to 92.5] | 93.0 [90.7 to 94.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.9576, Miettinen & Nurminen method — One-sided p-value based on Miettinen & Nurminen method stratified by prior docetaxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No) with small strata; Percent Difference = -2.7, 95% CI 2-sided [-5.8 to 0.4] — Percent difference and associated 95% CI were calculated using Miettinen & Nurminen method stratified by prior docetaxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No)

10. Secondary Outcome: Prostate-specific Antigen (PSA) Undetectable
Description: PSA undetectable rate was defined as the percentage of participants with detectable PSA (> 0.2 ng/mL) at baseline, which becomes undetectable (< 0.2 ng/mL) during study treatment.
Time Frame: Up to Approximately 32 Months
Population: All randomized participants with detectable PSA at baseline and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 587 | 585
Percentage of Participants | 63.4 [59.3 to 67.3] | 64.1 [60.1 to 68.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.6053, Miettinen & Nurminen — [p-value comment as in outcome 9, analysis 1]; Percent difference = -0.8, 95% CI 2-sided [-6.3 to 4.8] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Objective Response Rate (ORR) Per PCWG-Modified RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants with complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease (NED) on base scan per PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG).
Time Frame: Up to Approximately 32 Months
Population: All randomized participants with measurable disease at baseline and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 248 | 245
Percentage of Participants | 65.7 [59.5 to 71.6] | 71.8 [65.8 to 77.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide + ADT vs Placebo + Enzalutamide + ADT; Test type: Other; p = 0.9105, Miettinen & Nurminen — One-sided p-value based on Miettinen & Nurminen method stratified prior docataxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No) with small strata; Percent difference = -5.6, 95% CI 2-sided [-13.7 to 2.6] — Percent difference and associated 95% CI were calculated using Miettinen & Nurminen method stratified by prior docataxel for mHSPC (Yes/No) and presence of high-volume disease (Yes/No)

12. Secondary Outcome: Duration of Response (DOR) Per PCWG- Modified RECIST 1.1 as Assessed by BICR
Description: DOR was defined as the time from first documented evidence of complete response (CR) or partial response (PR) per PCWG and RECIST 1.1 criteria until progressive disease (PD) or death. PD per RECIST 1.1 was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of a least 5 mm. PD per PCWG was the appearance of >2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and were persistent for >6 weeks. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to Approximately 32 Months
Population: All randomized participants who demonstrated a CR or PR, and had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
Number analyzed (Participants) | 163 | 176
Months | NA [22.2 to NA] — NA = Median and upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response. | NA [NA to NA] — NA = Median, lower limit and upper limit of 95% CI for DOR cannot be calculated at the time of last disease assessment due to insufficient number of participants with response.

13. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Participants who experienced an AE will be reported for each arm.
Time Frame: Up to Approximately 59 Months
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported for each arm.
Time Frame: Up to Approximately 59 Months
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: Up to Approximately 32 months
Description: All-cause mortality was reported on all randomized participants and adverse events (serious and non-serious) were reported on all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded.
Arm/Group | Pembrolizumab + Enzalutamide + ADT | Placebo + Enzalutamide + ADT
All-Cause Mortality (participants affected / at risk) | 105/626 | 93/625
Serious Adverse Events (participants affected / at risk) | 252/625 | 145/625
Other Adverse Events (participants affected / at risk) | 588/625 | 551/625
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide + ADT (N=625) | Placebo + Enzalutamide + ADT (N=625)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 3 (3)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 7 (7) | 7 (7)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Normal tension glaucoma (Eye disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 7 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (9)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Sudden death (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 2 (3) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 5 (5) | 0 (0)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 6 (6)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Joint tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 7 (8)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (16) | 7 (7)
Urosepsis (Infections and infestations) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 0 (0)
Noninfective encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Progressive bulbar palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 3 (4) | 5 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 2 (3)
Device malfunction (Product Issues) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (2)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 3 (4)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Immunotactoid glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide + ADT (N=625) | Placebo + Enzalutamide + ADT (N=625)
Anaemia (Blood and lymphatic system disorders) | 97 (139) | 85 (108)
Hypothyroidism (Endocrine disorders) | 82 (82) | 25 (25)
Abdominal pain (Gastrointestinal disorders) | 32 (41) | 29 (33)
Constipation (Gastrointestinal disorders) | 108 (133) | 103 (117)
Diarrhoea (Gastrointestinal disorders) | 127 (196) | 73 (92)
Nausea (Gastrointestinal disorders) | 105 (125) | 75 (86)
Vomiting (Gastrointestinal disorders) | 35 (43) | 29 (36)
Asthenia (General disorders) | 80 (101) | 55 (66)
Fatigue (General disorders) | 194 (236) | 178 (200)
Oedema peripheral (General disorders) | 67 (73) | 50 (54)
Pyrexia (General disorders) | 63 (68) | 26 (31)
COVID-19 (Infections and infestations) | 75 (76) | 75 (76)
Urinary tract infection (Infections and infestations) | 37 (43) | 31 (40)
Fall (Injury, poisoning and procedural complications) | 44 (51) | 53 (64)
Alanine aminotransferase increased (Investigations) | 73 (89) | 38 (39)
Aspartate aminotransferase increased (Investigations) | 74 (93) | 39 (43)
Blood alkaline phosphatase increased (Investigations) | 40 (49) | 18 (20)
Blood creatinine increased (Investigations) | 36 (58) | 20 (29)
Weight decreased (Investigations) | 57 (62) | 20 (25)
Decreased appetite (Metabolism and nutrition disorders) | 91 (107) | 52 (59)
Hyperglycaemia (Metabolism and nutrition disorders) | 58 (90) | 51 (71)
Arthralgia (Musculoskeletal and connective tissue disorders) | 181 (251) | 161 (208)
Back pain (Musculoskeletal and connective tissue disorders) | 102 (114) | 113 (125)
Bone pain (Musculoskeletal and connective tissue disorders) | 39 (40) | 33 (36)
Myalgia (Musculoskeletal and connective tissue disorders) | 54 (63) | 50 (65)
Neck pain (Musculoskeletal and connective tissue disorders) | 32 (33) | 21 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 65 (81) | 66 (83)
Dizziness (Nervous system disorders) | 59 (66) | 46 (53)
Dysgeusia (Nervous system disorders) | 37 (39) | 23 (24)
Headache (Nervous system disorders) | 79 (98) | 65 (81)
Paraesthesia (Nervous system disorders) | 22 (28) | 41 (43)
Insomnia (Psychiatric disorders) | 62 (71) | 47 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (54) | 44 (51)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 (60) | 24 (25)
Dry skin (Skin and subcutaneous tissue disorders) | 49 (56) | 48 (55)
Pruritus (Skin and subcutaneous tissue disorders) | 110 (142) | 55 (73)
Rash (Skin and subcutaneous tissue disorders) | 148 (200) | 58 (66)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 56 (61) | 15 (23)
Hot flush (Vascular disorders) | 110 (119) | 144 (148)
Hypertension (Vascular disorders) | 108 (130) | 130 (155)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04191096/Prot_SAP_000.pdf